CLINICAL TRIAL: NCT00201279
Title: Phase III Placebo-Controlled Chemoprevention Study of Oral Cavity Squamous Cell Carcinoma Patients
Brief Title: Chemoprevention Study of Oral Cavity Squamous Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Changhua Christian Hospital (Other); China Medical University Hospital (Other); Buddhist Tzu Chi General Hospital (Other); Taichung Veterans General Hospital (Other); Mackay Memorial Hospital (Other); Chang Gung Memorial Hospital (Other); Koo Foundation Sun Yat-Sen Cancer Center (Other); Chi Mei Medical Hospital (Other); National Cheng-Kung University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: T1399
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-01

CONDITIONS: Oral Cavity; Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell

INTERVENTIONS:
Drug: 13-cis Retino Acid

SUMMARY:
The purpose of this study is to study the effect of 13-cis retinoic acid in preventing second primary malignancy in the oral cavity cancer patients after curative local treatment and to study the toxicity and compliance of 13-cis retinoic acid.

DETAILED DESCRIPTION:
There are more than one thousand deaths annually from head and neck cancer in Taiwan (excluding nasopharyngeal carcinoma) and the majority of treatment failures are related to recurrence of primary disease. Only patients with early-stage disease have high cure rates, but they remain at risk for the development of second primary tumors.

Second primary malignancies occur at a constant annual rate of 5% to 7% in all head and neck cancer patients1. Furthermore, because the mortality from primary disease recurrence plateaus after 2 to 3 years in patients with locally advanced disease, second primary tumors become the major cause of late cancer mortality.

Sporn et al defined chemoprevention as an effort to arrest or reverse premalignant cells during their progression to invasive malignancy2,3. The concept of chemoprevention has evolved to include the use of specific compounds, rather than general dietary changes, to prevent the development of cancer.

Hong et al studied the effects of 13-cis retinoic acid on patients with history of head and neck cancers 4. After treatment of head and neck primary cancers with either radiotherapy or surgery or both, 103 patients were randomized to receive either adjuvant 13-cis retinoic acid or placebo. In an update of this trial with 55 months of follow-up, 16 patients (31%) in the placebo group had developed second primary tumors, whereas 7 patients (14%) in the treatment group had developed second primary tumors (p=0.04) 5. Betel quid chewing becomes increasingly popular in Taiwan. Exposure to both smoking and betel quid significantly increases the risk of oral cavity cancer6. The hazard of developing second primary tumors is high in this population, therefore, chemoprevention is worthy of trial.

Use of 13-cis RA for chemoprevention of head and neck cancer only has been published by Hong et al. Their cases included a variety of head and neck cancers that are known to be not a homogenous group. The risk of second primary is different for different primary sites. Therefore, the value of 13-cis RA in chemoprevention is not conclusively addressed. In our proposal, only oral cavity cancer is included and the result will be more convincing. The result could be the basis of further chemoprevention clinical trial or guideline for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinically free of disease after having undergone surgery for histologically confirmed primary SCC of the oral cavity(Buccal mucosa +Oral tongue )
* Without any risk factor of recurrence listed below:
* Nodal extracapsular spread of disease (ECS)
* Number of positive node > 2
* Perineural involvement
* Lymphovascular emboli/permeation in resected surgical specimen
* Histologically positive surgical margins, but no gross residual disease

Exclusion Criteria:

* A KPS of less than 50 percent
* Serum creatinine and/or GOT/GPT greater than 2 times upper normal limit
* Distant metastasis
* Has previously received chemotherapy
* Has received within the two years diagnosis of any cancer
* Women of reproductive capacity
* Cases beyond the age range of 20-65 years.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342
Dates: Start 1999-04; Study Completion 2012-09

PRIMARY OUTCOMES:
Primary tumor recurrence

SECONDARY OUTCOMES:
The development of a second primary tumor

CONTACTS AND LOCATIONS:
Overall Officials: Mow-Ming Hsu, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- See also: Related Info — http://www.nhri.org.tw